CLINICAL TRIAL: NCT02025205
Title: A Multicentre, Prospective, Randomized, Controlled, One-way Crossover Investigation of Endobronchial Valve (EBV) Therapy vs. Standard of Care (SoC) in Homogeneous Emphysema
Brief Title: Improving Patient Outcomes by Selective Implantation of the Zephyr EBV - Study
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulmonx International Sàrl (Industry)
Responsible Party: Sponsor
Organization: Pulmonx Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 630-0014
Record Dates: First submitted 2013-12-21; First posted 2013-12-31 (Estimated); Results first posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-07

CONDITIONS: COPD Patients With Homogeneous Emphysema; Endoscopic Lung Volume Reduction With Endobronchial Valve

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ELVR with Endobronchial Valves (Experimental): Endoscopic Lung Volume Reduction with Zephyr Endobronchial Valve
  Interventions: Device: Endobronchial Valve
- Standard of Care (No Intervention): Patients will receive optimal drug therapy and medical management according to clinical practice.

INTERVENTIONS:
Device: Endobronchial Valve — Endoscopic Lung Volume Reduction with Zephyr Endobronchial Valve
  Arms: ELVR with Endobronchial Valves

SUMMARY:
The aim of this prospective, randomized, controlled, one-way crossover study is to assess and compare the efficacy of the Zephyr endobronchial valves vs. Standard of Care (SoC) in patients suffering from COPD with Homogeneous Emphysema. Patients will be followed up for 12 months after randomization. Patients in the SoC arm will crossover to the EBV treatment arm after the 6-month visit and will be followed up for 6 additional months.The primary objective is the variation of FEV1 between baseline and 3-month follow-up visit. The secondary objectives will evaluate quality of life, exercise capacity, dyspnea (including BODE index) changes, target lobe volume reduction, as well as safety outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Homogeneous emphysema
* 15% ≤ FEV1 ≤ 45% predicted
* TLC > 100% predicted
* RV ≥ 200% predicted
* 6MWT ≥ 150 m
* Non-smoker > 8 weeks prior to study entry
* Absence of Collateral Ventilation in the target lobe

Exclusion Criteria:

* Active pulmonary infection
* More than 3 exacerbations with hospitalizations over the past 12 months
* Pulmonary hypertension (sPAP > 45 mmHg)
* MI or other relevant CV events in the past 6 months
* Alpha-1 antitrypsin deficiency
* Bronchiectasis
* Prior LVR or LVRS procedure
* > 20% difference in perfusion between right and left lung
* Hypercapnia (paCO2 > 55 mmHg
* Asthma
* Use of more than 25 mg/day prednisolone or equivalent
* Severe bullous emphysema
* Systemic or malignant disease with high death probability within 12 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arschang Valipour, MD, PhD, FCCP, Principal Investigator — Ludwig-Boltzmann-Institute for COPD and Respiratory Epidemiology Otto-Wagner-Spital 1140 Wien / Austria; Felix Herth (co-principal investigator), MD, Principal Investigator — Heidelberg University; Ralf Eberhardt (co-principal investigator), MD, Principal Investigator — Heidelberg University
Locations (8):
- Ludwig-Boltzmann-Institut für COPD und Pneumologische Epidemiologie, Vienna, Austria
- Germany (6):
  - Charité Campus Virchow-Klinikum, Berlin
  - Ruhrlandklinik, Westdeutsches Lungenzentrum, Essen
  - Lungenabteilung Thoraxzentrum Hamburg, Hamburg
  - Thoraxklinik am Universitäts klinikum Heidelberg, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Klinikum Nürnberg Nord, Nuremberg
- Department of pulmonary dieases, University Medical Center, Groningen, Netherlands

REFERENCES:
- [Derived] Bakker JT, Hartman JE, Klooster K, Charbonnier JP, Tsiaousis M, Vliegenthart R, Slebos DJ. Endobronchial valve treatment improves chest-CT diaphragm configuration in COPD. Respir Med. 2024 Nov-Dec;234:107856. doi: 10.1016/j.rmed.2024.107856. Epub 2024 Nov 6. PMID 39515624

RESULTS

PARTICIPANT FLOW:
Groups:
- BLVR With Zephyr Endobronchial Valves: Bronchoscopic Lung Volume Reduction with Zephyr Endobronchial Valves
  Endobronchial Valve: Bronchoscopic Lung Volume Reduction (BLVR) with Zephyr Endobronchial Valve
Period: Overall Study
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Started | 43 | 50
Completed | 40 | 47
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ELVR With Endobronchial Valves | Standard of Care | Total
Number analyzed (Participants) | 43 | 50 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (6.3) | 63.2 (6.0) | 63.7 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 34 | 57
  Male | 20 | 16 | 36
Region of Enrollment [Number; unit: participants]
  Netherlands | 9 | 14 | 23
  Austria | 8 | 13 | 21
  Germany | 26 | 23 | 49
Height [Mean (Standard Deviation); unit: cm] | 168.7 (10.0) | 165.4 (9.1) | 166.9 (9.6)
Weight [Mean (Standard Deviation); unit: kg] | 67.9 (15.4) | 62.2 (12) | 64.8 (13.9)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.7 (4.3) | 22.6 (3.7) | 23.1 (4.0)
Pack Years Smoking History [Median (Standard Deviation); unit: pack-years] — Population: The number of subjects in the EBV and SoC group analyzed for Pack year smoking history is less than the overall population, due to missing data.
  pack-years
    number analyzed (Participants) | 41 | 48 | 89
    (all) | 41.5 (19.6) | 42.5 (22.0) | 42.0 (20.8)
Gold stage [Count of Participants; unit: Participants] — The GOLD system uses the term "stages" to refer to the different levels of COPD. Participants graded as GOLD Stage III are considered to have Severe COPD. Participants graded as GOLD Stage IV are considered to have Very Severe COPD.
  Participants
    Gold Stage III | 18 | 23 | 41
    Gold Stage IV | 25 | 27 | 52
Emphysema score [Mean (Standard Deviation); unit: percent] — Emphysema score was assessed as the percentage of voxels of less than -910 Hounsfield units on Computerized Tomography (CT). Scores range from 0 to 100%, with higher scores indicating more emphysematous destruction.
  percent | 68.0 (7.5) | 65.8 (6.9) | 66.8 (7.3)
Heterogeneity index [Mean (Standard Deviation); unit: units on a scale] — Difference in emphysema destruction scores between potential target and ipsilateral lung lobes, calculated from the high-resolution computer tomography scan (HRCT) read. The classification of Homogeneous or Heterogeneous emphysema follows the below criteria:
  1. Homogeneous emphysema = heterogeneity index between target and adjacent lobes of <15%.
  2. Heterogeneous emphysema = heterogeneity index between target and adjacent lobes of ≥15%.
  units on a scale | 6.8 (5.7) | 5.0 (6.3) | 5.9 (6.0)
FEV1 (liters) [Mean (Standard Deviation); unit: Liters] | 0.8 (0.2) | 0.8 (0.2) | 0.8 (0.2)
FEV1 (% predicted) [Mean (Standard Deviation); unit: % predicted] | 28.4 (6.3) | 30.0 (6.6) | 29.3 (6.5)
Residual Volume (RV) (Liters) [Mean (Standard Deviation); unit: Liters] | 5.7 (1.1) | 5.2 (1.2) | 5.5 (1.2)
Residual Volume (RV) (% predicted) [Mean (Standard Deviation); unit: % predicted] | 277.3 (55.2) | 273.7 (63.4) | 275.4 (59.4)
Total Lung Capacity (TLC) (Liters) [Mean (Standard Deviation); unit: Liter] | 8.4 (1.6) | 7.6 (1.4) | 8.0 (1.5)
Total Lung Capacity (TLC) (% predicted) [Mean (Standard Deviation); unit: % predicted] | 144.9 (21.2) | 144.2 (17.6) | 144.6 (19.3)
FEV1/FVC (%) [Mean (Standard Deviation); unit: percent] | 36.3 (7.2) | 35.8 (8.6) | 36.0 (7.9)
RV/TLC (%) [Mean (Standard Deviation); unit: percent] | 69.0 (6.3) | 68.2 (7.1) | 68.6 (6.7)
6 Minute Walk Distance (meters) [Mean (Standard Deviation); unit: meters] | 308.0 (91.3) | 328.3 (92.6) | 318.9 (92.1)
SGRQ Total Score [Mean (Standard Deviation); unit: points on a scale] — The St. George's Respiratory Questionnaire measures health status (quality of life) in patients with diseases of airways obstruction. The questionnaire comprises of two parts:
  Part I: Symptoms (frequency & severity) Part II: Activities that cause or are limited by breathlessness; Impacts (social functioning, psychological disturbances resulting from airways disease)
  A Total score is calculated which summarizes the impact of the disease on overall health status. Scores range from 0 to 100, with higher scores indicating more limitations. Population: The number of subjects in the EBV and SoC group analyzed for SGRQ Total Score is less than the overall population, due to missing data.
  points on a scale
    number analyzed (Participants) | 41 | 49 | 90
    (all) | 63.2 (13.7) | 59.3 (15.6) | 61.1 (14.8)
The COPD Assessment Test (CAT) total score (derived) [Mean (Standard Deviation); unit: points on a scale] — The COPD Assessment Test (CAT) is an eight-item questionnaire designed to quantify the impact of COPD symptoms on the health status of patients. The CAT provides a score of 0-40 to indicate the impact of disease. Higher scores denote a more severe impact of COPD on a patient's life. Population: The number of subjects in the SoC group analyzed for CAT Total Score, derived is less than the overall population, due to missing data.
  points on a scale
    number analyzed (Participants) | 43 | 49 | 92
    (all) | 23.4 (6.8) | 22.8 (6.0) | 23.1 (6.3)
EQ-5D Summary Index [Mean (Standard Deviation); unit: points on a scale] — EQ-5D is a standardized instrument to measure health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5D consists of a descriptive system and the EQ VAS.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-5D health states may be converted into a single summary index by applying a formula that attaches weights to each of the levels in each dimension. The maximum score of 1 indicates the best health state, while 0 indicates the worst health state. Population: The number of subjects in the EBV and SoC group analyzed for EQ-5D summary index, Europe is less than the overall population, due to missing data.
  points on a scale
    number analyzed (Participants) | 39 | 48 | 87
    (all) | 0.5 (0.3) | 0.6 (0.2) | 0.6 (0.3)
EQ-5D health state today [Mean (Standard Deviation); unit: score] — EQ-5D is a standardized instrument to measure health-related quality of life. The EQ-5D consists of a descriptive system and the EQ VAS (visual analogue scale). The EQ VAS corresponds to the EQ-5D health state today and records the respondent's self-rated health on a vertical scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
  Scores range from 0 to 100, with lower scores indicating worse health states. Population: The number of subjects in the EBV and SoC group analyzed for EQ-5D Health State today is less than the overall population, due to missing data.
  score
    number analyzed (Participants) | 41 | 48 | 89
    (all) | 40.3 (14.4) | 49.3 (19.3) | 45.2 (17.7)
mMRC Dyspnea Grade score [Mean (Standard Deviation); unit: points on a scale] — The mMRC (Modified Medical Research Council) stratifies severity of dyspnea in respiratory diseases. The severity of dyspnea is rated on a scale of 0 to 4, with higher scores indicating more limitations. Population: The number of subjects in the EBV group analyzed for mMRC breathlessness grade is less than the overall population, due to missing data.
  points on a scale
    number analyzed (Participants) | 42 | 50 | 92
    (all) | 2.7 (0.8) | 2.4 (1.0) | 2.5 (0.9)
BODE index [Mean (Standard Deviation); unit: points on a scale] — The BODE Index is comprised of a person's body mass index ("B"), airway obstruction ("O"), dyspnea ("D"), and exercise tolerance ("E"). Each of these components is graded on a scale of either 0 to 1 or 0 to 3. The final value-ranging from 0 to 10-provides doctors a percentage of how likely a person is to survive for four years. The final BODE tabulation is described as follows:
  0 to 2 points: 80 percent likelihood of survival 3 to 4 points: 67 percent likelihood of survival 5 of 6 points: 57 percent likelihood of survival 7 to 10 points: 18 percent likelihood of survival Population: The number of subjects in the EBV group analyzed for BODE index is less than the overall population, due to missing data.
  points on a scale
    number analyzed (Participants) | 42 | 50 | 92
    (all) | 5.7 (1.4) | 5.2 (1.7) | 5.4 (1.6)
EQ-5D Mobility [Count of Participants; unit: Participants] — Population: The number of subjects in the EBV and SOC group analyzed for EQ-5D mobility is less than the overall population, due to missing data.
  Participants
    number analyzed (Participants) | 41 | 48 | 89
    No problems | 8 | 15 | 23
    Some problems | 32 | 33 | 65
    Confined to bed | 1 | 0 | 1
EQ-5D Self-Care [Count of Participants; unit: Participants] — Population: The number of subjects in the EBV and SoC group analyzed for EQ-5D Self-Care is less than the overall population, due to missing data.
  Participants
    number analyzed (Participants) | 41 | 48 | 89
    No problems | 13 | 27 | 40
    Some problems | 25 | 21 | 46
    Unable | 3 | 0 | 3
EQ-5D usual activities [Count of Participants; unit: Participants] — Population: The number of subjects in the EBV and SoC group analyzed for EQ-5D Usual Activities is less than the overall population, due to missing data.
  Participants
    number analyzed (Participants) | 41 | 48 | 89
    No problems | 2 | 5 | 7
    Some problems | 32 | 32 | 64
    Unable | 7 | 11 | 18
EQ-5D Pain/Discomfort [Count of Participants; unit: Participants] — Population: The number of subjects in the EBV and SoC group analyzed for EQ-5D pain/discomfort is less than the overall population, due to missing data.
  Participants
    number analyzed (Participants) | 39 | 48 | 87
    No | 16 | 28 | 44
    Moderate | 20 | 16 | 36
    Extreme | 3 | 4 | 7
EQ-5D Anxiety/Depression [Count of Participants; unit: Participants] — Population: The number of subjects in the EBV and SoC group analyzed for EQ-5D anxiety/depression is less than the overall population, due to missing data.
  Participants
    number analyzed (Participants) | 41 | 48 | 89
    No | 16 | 22 | 38
    Moderate | 16 | 24 | 40
    Extreme | 9 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Forced Expiratory Volume in 1 s (FEV1) (ITT Population)
Description: Percentage change in FEV1 at 3 months relative to Baseline in the EBV group, compared to the SoC group.
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 43 | 50
percent change | 13.7 (28.2) | -3.2 (13)

2. Secondary Outcome: Absolute Change in Target Lobe Volume for EBV Group (ITT Population)
Description: Target Lobe Volume Reduction (TLVR) was evaluated by quantitative analysis of HRCT scans at Baseline and at 3-months post-valve placement to measure the target lobe volume.
Time Frame: At baseline and after 3 months
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | BLVR With Zephyr Endobronchial Valves
Number analyzed (Participants) | 36
mL | 1195 (683.2)

3. Secondary Outcome: Percent Change in Target Lobe Volume for EBV Group (ITT Population)
Description: as for outcome 2
Time Frame: At baseline and after 3 months
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | BLVR With Zephyr Endobronchial Valves
Number analyzed (Participants) | 36
Percent change | 64.9 (32.5)

4. Secondary Outcome: Percent of Subjects in the EBV Group With a Target Lobe Volume Reduction (TLVR) of ≥ 350ml at 3 Months
Description: The threshold of TLVR ≥350 mL was used to determine the proportion of subjects that achieved this amount of TLVR in the EBV group.
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | BLVR With Zephyr Endobronchial Valves
Number analyzed (Participants) | 36
Participants
  Yes | 32
  No | 4

5. Secondary Outcome: Absolute Change in FEV1 (L) Post Bronchodilator at 3 Months
Description: The mean absolute change in FEV1(L) relative to Baseline at 3 months between the EBV and SoC groups
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 43 | 50
liters | 0.1 (0.2) | -0.02 (0.1)

6. Secondary Outcome: Absolute Change in FEV1 (% Predicted) Post Bronchodilator at 3 Months
Description: The mean absolute change in FEV1(% Predicted) relative to Baseline at 3 months between the EBV and SoC groups
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percent predicted
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 43 | 50
Percent predicted | 3.4 (6.5) | -1.3 (4.2)

7. Secondary Outcome: Absolute Change in Residual Volume (RV) at 3 Months
Description: Mean absolute change in Residual Volume relative to Baseline at 3 months between the EBV and SoC groups
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 43 | 50
liters | -0.4 (0.9) | 0.1 (0.9)

8. Secondary Outcome: Percent Change in Residual Volume (RV) at 3 Months
Description: Mean percent change in Residual Volume relative to Baseline at 3 months between the EBV and SoC groups
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 43 | 50
Percent change | -6.7 (13.6) | 2.7 (19.0)

9. Secondary Outcome: Percent Predicted Change in Residual Volume at 3 Months
Description: Percent predicted change in RV relative to Baseline at 3 months between the EBV and SoC groups
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 43 | 50
Percent change | -21.1 (47.6) | -0.3 (53.6)

10. Secondary Outcome: Absolute Change in Six-Minute Walk Distance at 3 Months
Description: Mean absolute change in the 6MWD from Baseline to 3 months in the EBV group compared to the SOC
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 42 | 50
meters | 22.6 (66.6) | -17.3 (52.8)

11. Secondary Outcome: Percent Change in Six-Minute Walk Distance at 3 Months
Description: Mean percent change in the 6MWD from Baseline to 3 months in the EBV group compared to the SOC
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 42 | 50
Percent change | 10.6 (26.5) | -3.9 (18.0)

12. Secondary Outcome: Absolute Change in the SGRQ Total Score From Baseline to 3 Months
Description: Mean absolute change in the St. George's Respiratory Questionnaire Total Score from Baseline to 3 months in the EBV group compared to the SoC group. Scores range from 0 to 100, with higher scores indicating more limitations.
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 37 | 48
points on a scale | -8.6 (11.3) | 1.0 (9.4)

13. Secondary Outcome: Percent Change (%) in the SGRQ Total Score From Baseline to 3 Months
Description: Mean percent change in the SGRQ Total Score from Baseline to 3 months in the EBV group compared to the SoC group
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 37 | 48
percent change | -14.8 (19.5) | 3.9 (20.5)

14. Secondary Outcome: Absolute Change in the mMRC Dyspnea Score From Baseline to 3 Months
Description: Mean absolute change in the Modified Medical Research Council (mMRC) Dyspnea Score from Baseline to 3 months in the EBV group compared to the SoC group. The mMRC (Modified Medical Research Council) stratifies severity of dyspnea in respiratory diseases. The severity of dyspnea is rated on a scale of 0 to 4, with higher scores indicating more limitations.
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 41 | 50
points on a scale | -0.4 (1.0) | 0.2 (1.0)

15. Secondary Outcome: Percent Change (%) in the mMRC Dyspnea Score From Baseline to 3 Months
Description: Mean percent change in the mMRC Dyspnea Score from Baseline to 3 months in the EBV group compared to the SoC group. The mMRC (Modified Medical Research Council) stratifies severity of dyspnea in respiratory diseases. The severity of dyspnea is rated on a scale of 0 to 4, with higher scores indicating more limitations.
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 41 | 49
Percent change | -11.0 (40.0) | 14.3 (59.3)

16. Secondary Outcome: Absolute Change in the CAT Total Score From Baseline to 3 Months
Description: Mean absolute change in the COPD Assessment Test (CAT) Total Score from Baseline to 3 months in the EBV group compared to the SoC group.
  The COPD Assessment Test (CAT) is an eight-item questionnaire designed to quantify the impact of COPD symptoms on the health status of patients. The CAT provides a score of 0-40 to indicate the impact of disease.
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 42 | 49
points on a scale | -1.5 (5.6) | -0.7 (3.7)

17. Secondary Outcome: Percent Change (%) in CAT Total Score From Baseline to 3 Months
Description: The COPD Assessment Test (CAT) is an eight-item questionnaire designed to quantify the impact of COPD symptoms on the health status of patients. The CAT provides a score of 0-40 to indicate the impact of disease. Higher scores denote a more severe impact of COPD on a patient's life.
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 42 | 49
percent change | -4.9 (30.2) | -0.9 (16.5)

18. Secondary Outcome: Absolute Change in EQ-5D Summary Index From Baseline to 3 Months
Description: Mean absolute change in the EQ-5D Summary Index from Baseline to 3 months in the EBV group compared to the SoC group.
  EQ-5D is a standardized instrument to measure health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5D consists of a descriptive system and the EQ VAS.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-5D health states may be converted into a single summary index by applying a formula that attaches weights to each of the levels in each dimension. The maximum score of 1 indicates the best health state, while 0 indicates the worst health state.
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 39 | 48
points on a scale | 0.1 (0.2) | 0.01 (0.2)

19. Secondary Outcome: Percent Change (%) in EQ-5D Summary Index From Baseline to 3 Months
Description: Mean percent change in EQ-5D Summary Index from Baseline to 3 months in the EBV group compared to the SoC group.
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 39 | 48
percent change | 32.7 (70.1) | 26.2 (115.0)

20. Secondary Outcome: Absolute Change in EQ-5D VAS (Health State Today) Score From Baseline to 3 Months
Description: Mean absolute change in the EQ-5D VAS (Health State Today) Score from Baseline to 3 months in the EBV group compared to the SoC group. Scores range from 0 to 100, with higher scores indicating better outcome.
Time Frame: At baseline and after 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Number analyzed (Participants) | 41 | 48
points on a scale | 12.7 (17.7) | -0.4 (17.6)

ADVERSE EVENTS:
Arm/Group | BLVR With Zephyr Endobronchial Valves | Standard of Care
Serious Adverse Events (participants affected / at risk) | 28/43 | 16/50
Other Adverse Events (participants affected / at risk) | 30/43 | 22/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLVR With Zephyr Endobronchial Valves (N=43) | Standard of Care (N=50)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 13 (19) | 12 (12)
Diagnostic bronchoscopy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLVR With Zephyr Endobronchial Valves (N=43) | Standard of Care (N=50)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Insomnia (Nervous system disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 14 (25) | 10 (14)
Common cold (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 6 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Mucus production (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary granulations (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary infection (Infections and infestations) | 3 (4) | 0 (0)
Pulmonary shunt (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Thoracic pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pulmonary lesion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No